CLINICAL TRIAL: NCT05584423
Title: The Correlation Between the Difficulty of Colonoscopy and the Patient's Personality
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-DCPP
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-05

CONDITIONS: Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore the correlation between the difficulty of colonoscopy and the patients' personality in the population receiving initial colonoscopy in Peking Union Medical College Hospital. The main question it aims to answer is: Whether the difficulty of colonoscopy is related to any personality score of big five personality dimensions

Participants will:

1. Receive routine colonoscopy
2. Fill out the GAD-7 and PHQ-9 scales
3. Fill out the Big Five Personality Questionnaire.

DETAILED DESCRIPTION:
Colonoscopy as an invasive test may cause pain, discomfort and anxiety to the patient . Insertion time and patient pain scores are indicators of the degree of colonoscopy difficulty, with the incidence of difficult colonoscopy being approximately 25% . It is usually defined as a difficult colonoscopy when the insertion time is more than 10 minutes. Several studies have shown that certain risk factors can help us predict the occurrence of difficult colonoscopy, such as gender, age, BMI, bowel preparation, and history of abdominal or pelvic surgery .

In addition to the objective factors mentioned above, the patient's personality, mood and psychological state may also have an impact on the difficulty of colonoscopy. In clinical practice, endoscopists have observed that patients with anxiety-prone or obsessive personalities tend to have a higher incidence of difficult colonoscopies, but few studies have explored the predictive role of patient personality on the degree of difficulty in colonoscopy. In addition, because personality stability may be influenced by anxiety and depression levels as well as specific strong situations, the patient's recent anxiety and depression levels should also be taken into account. We therefore used the Generalized Anxiety Scale (GAD-7) and the 9-item Patient Health Questionnaire Depression Scale (PHQ-9) to assess patients' recent levels of anxiety and depression, respectively.

The Big Five is currently recognized as the most comprehensive model of personality analysis and has been widely used in clinical and scientific research. The Big Five includes extraversion、extraversion、conscientiousness、neuroticism、openness. This study intends to use the Chinese version of the Big Five Personality Questionnaire to test the scores of patients in the five personality dimensions, in order to observe whether the difficulty of colonoscopy is related to the scores of any personality dimension.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Patients or family members were able to understand the study protocol and willing to participate in this study by signing informed consent.
3. Those who underwent colonoscopy at the Gastrointestinal Endoscopy Center of Peking Union Medical College Hospital.

Exclusion Criteria:

1. Patients who have taken colonoscopy before
2. Patients who are unable to read or write
3. Patients with severe mental disorders, organic brain mental disorders
4. those with poor bowel preparation (BBPS < 6 )
5. patients with chronic constipation, history of intestinal diverticula
6. Patients who have undergone previous colorectal surgery
7. those with previous findings of severe colonic strictures or obstructive tumors
8. patients who are pregnant or breastfeeding
9. patients with severe infectious diseases.
10. Patients with inflammatory bowel disease, familial polyposis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who meet the eligibility criteria and undergo colonoscopy at Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
insertion time | During colonoscopy procedure
  Total time from the insertion of the colonoscope into the anus until the colonoscope reaches the cecum

SECONDARY OUTCOMES:
pain scores | colonoscopy procedure
  The degree of maximum abdominal pain
Willingness to undergo colonoscopy again questionnaire | colonoscopy procedure
  After colonoscopy, ask the patient if they are willing to accept colonoscopy again if they have the same chief complaint

CONTACTS AND LOCATIONS:
Overall Officials: DONG WU, M.D., Principal Investigator — Peking Union Medical College Hospital; SHENGYU ZHANG, Study Director — Peking Union Medical College Hospital; YINAN JIANG, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Bond JH, Winawer S, Levin TR, Burt RW, Johnson DA, Kirk LM, Litlin S, Lieberman DA, Waye JD, Church J, Marshall JB, Riddell RH; U.S. Multi-Society Task Force on Colorectal Cancer. Quality in the technical performance of colonoscopy and the continuous quality improvement process for colonoscopy: recommendations of the U.S. Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2002 Jun;97(6):1296-308. doi: 10.1111/j.1572-0241.2002.05812.x. No abstract available. PMID 12094842
- [Background] van Doorn SC, van Vliet J, Fockens P, Dekker E. A novel colonoscopy reporting system enabling quality assurance. Endoscopy. 2014 Mar;46(3):181-7. doi: 10.1055/s-0034-1364877. Epub 2014 Feb 5. PMID 24500977
- [Background] Ersoz F, Toros AB, Aydogan G, Bektas H, Ozcan O, Arikan S. Assessment of anxiety levels in patients during elective upper gastrointestinal endoscopy and colonoscopy. Turk J Gastroenterol. 2010 Mar;21(1):29-33. doi: 10.4318/tjg.2010.0044. PMID 20533109
- [Background] Hull T, Church JM. Colonoscopy--how difficult, how painful? Surg Endosc. 1994 Jul;8(7):784-7. doi: 10.1007/BF00593441. PMID 7974107
- [Background] Chung YW, Han DS, Yoo KS, Park CK. Patient factors predictive of pain and difficulty during sedation-free colonoscopy: a prospective study in Korea. Dig Liver Dis. 2007 Sep;39(9):872-6. doi: 10.1016/j.dld.2007.04.019. Epub 2007 Jul 24. PMID 17652041
- [Background] Jia H, Wang L, Luo H, Yao S, Wang X, Zhang L, Huang R, Liu Z, Kang X, Pan Y, Guo X. Difficult colonoscopy score identifies the difficult patients undergoing unsedated colonoscopy. BMC Gastroenterol. 2015 Apr 9;15:46. doi: 10.1186/s12876-015-0273-7. PMID 25886845
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Samuel DB, Widiger TA. A meta-analytic review of the relationships between the five-factor model and DSM-IV-TR personality disorders: a facet level analysis. Clin Psychol Rev. 2008 Dec;28(8):1326-42. doi: 10.1016/j.cpr.2008.07.002. Epub 2008 Jul 4. PMID 18708274
- [Derived] Wang D, Zhang S, Jiang Y, Ren Y, Kuai D, Zhao R, Wu D. Correlation between colonoscopy difficulty and personality traits: study protocol for a prospective, observational, multicentre study. BMJ Open. 2024 Dec 2;14(12):e090606. doi: 10.1136/bmjopen-2024-090606. PMID 39622570